CLINICAL TRIAL: NCT04010968
Title: Evaluation of Risk-Adapted and MRD-Driven Strategy for Untreated Fit Patients With Intermediate Risk Chronic Lymphocytic Leukemia: a Randomized Phase II Trial Comparing FCR and a Chemo-free Combination of Venetoclax and Ibrutinib. A FILO Study
Brief Title: Evaluation of Risk-Adapted and MRD-Driven Strategy for Untreated Fit Patients With Intermediate Risk Chronic Lymphocytic Leukemia
Acronym: ERADIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: AbbVie (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FILOCLL08 - ERADIC
Record Dates: First submitted 2019-06-20; First posted 2019-07-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Intermediate Risk Chronic Lymphocytic Leukemia; Fit Patients; Risk-Adapted and MRD-Driven Strategy
MeSH Terms: interventions — venetoclax; ibrutinib

STUDY DESIGN:
Intervention Model Description: Direct comparison between immuno-chemotherapy and effective chemo-free arm combining a BTK inhibitor and a Bcl2 inhibitor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCR (Active Comparator): FCR :
  * rituximab (R): 375 mg/m² IV D1 cycle 1 and 500 mg/m² IV D1 cycles 2 to 6.
  * fludarabine (F): 40 mg/m² orally, D2 to D4 - cycles 1 to 6.
  * cyclophosphamide (C): 250 mg/m² orally, D2 to D4 - cycles 1 to 6.
  Interventions: Drug: FCR
- venetoclax and ibrutinib (I+VEN) (Experimental): * ibrutinib: 420 mg/d orally, continuously from Month 1 to the end of treatment, either Month 15 or Month 27
  * venetoclax: stepwise weekly dose ramp-up beginning at Month 4 from a starting dose of 20 mg/d to the final dose of 400 mg/d (20, 50, 100, 200 and then 400 mg) over a 5 weeks, and then 400 mg/d continuously from Month 5 to the end of treatment, either Month 15 or Month 27.
  Interventions: Drug: venetoclax and ibrutinib (I+VEN)

INTERVENTIONS:
Drug: venetoclax and ibrutinib (I+VEN) — The treatment will start with ibrutinib alone for 3 months (lead-in phase) from Month 1 to Month 3 and then venetoclax will be added from Month 4 with an initial ramp-up period.
  The total duration of treatment with (I+VEN) will depend on the response achieved at Month 9:
  * if BM MRD at M9 < 0.01%, the treatment with (I+VEN) will be continued for 6 additional months until Month 15 and stopped then. MRD will be assessed at Month 15 (PB), Month 21 (PB) and Month 27 (PB and BM)
  * if BM MRD at M9 ≥ 0.01%, the treatment with (I+VEN) will be continued for 18 additional months until Month 27 and stopped then, whatever the results of MRD assessments that will be performed at the same time points as above.
  Arms: venetoclax and ibrutinib (I+VEN)
Drug: FCR — All patients will receive 6 cycles of FCR administered at 4 weeks intervals (D1 = D29) from Month 1 to Month 6.
  6 cycles of FCR will be administered at 4 weeks intervals (D1 = D29) from Month 1 to Month 6.
  Arms: FCR

SUMMARY:
The aim of this study is to test the potential benefit of an innovative combination of targeted therapy over the standard the immunochemotherapy (FCR). The interest in this study resides in an MRD driven discontinuation of the novel agents, and a fixed maximum duration of these agents. This design allows a true comparison of the efficacy of IV with the immuno-chemotherapy at 2 years of treatment and later.

Finally, other trials propose to include to all risk categories of patients, and we are developing here a stratification preventing the dilution of the results. The intermediate risk patients are the ones for which alternative to chemotherapy is critical, as chemotherapy is likely to alter the clonal evolution of their disease, whereas the low risk patients are already doing well with standard treatment and are likely to benefit from other therapies as well. The high risk patients, id est patients with 17p deletion and or TP 53 mutational status responded very well to new drugs as BTK inhibitors or BLC2 inhibitors.

DETAILED DESCRIPTION:
The combination of venetoclax (V) and ibrutinib (I) has recently emerged as a very effective therapy in both relapse and front-line settings. The preliminary results of the CLARITY (R/R CLL) and CAPTIVATE (untreated CLL) studies have demonstrated the promising potential of the I+VEN combination, which led to a very high rate of bone marrow MRD negativity. Moreover, the I+VEN combination might be given for only a definite period of time, contrarily to each of the two drugs which are given until disease progression or unacceptable toxicity per Smpc, according to their respective labels. The combination of V and I makes sense because of their in vitro synergy, non-overlapping toxicities and differential activity on different compartments of the disease. Therefore, the direct comparison in the front-line setting of the gold standard immuno-chemotherapy combining Rituximab plus Fludarabine and Cyclophosphamide FCR and an innovative chemo-free regimen combining I and V is essential in the intermediate-risk patients who benefit much less from FCR than the low-risk patients.

Primary objective : to evaluate the efficacy of the chemo-free combination of ibrutinib and venetoclax in previously untreated intermediate-risk CLL in a face to face comparison with the gold standard immuno-chemotherapy regimen FCR in order to assess if it may replace chemotherapy.

Secondary objectives :

* To determine the progression-free survival (PFS), event-free survival (EFS), overall survival (OS) and time to next treatment (TTNT)
* To evaluate the safety of the combination I + VEN
* To evaluate the dose intensity (RDI) of both treatments
* To assess the response (Complete Response / CR, CR with incomplete blood count recovery / CRi , CR with undetectable Measurable Residual Disease/MRD, Partial Remission / PR, nPR, with and without undetectable MRD)
* To determine the incidence of Richter transformation.

Innovative aspects of this trial

• Patient stratification based on robust prognostic factors. The risk stratification is based on IGHV status, genetic alterations by FISH analysis, karyotype and NGS (TP53 mutation), as now recommended by the IWCLL 2018 guidelines.

Focus on the intermediate-risk CLL patients (as defined above) who represent more than half of the CLL patients in need of first-line therapy and for whom replacement of FCR with a more effective innovative approach is a crucial issue.

* Direct comparison between immuno-chemotherapy and a very effective chemo-free arm combining a BTK inhibitor and a Bcl2 inhibitor.
* MRD use to optimize treatment strategy in the experimental arm. Early treatment discontinuation will be considered in patients who will rapidly reach bone marrow MRD negativity (< 10-4).
* Evaluation of a fixed duration of treatment with targeted therapy that will not be continued beyond 24 months
* Evaluation of the kinetics of reappearance of the disease by regular monitoring of the MRD in both arms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Immunophenotypically confirmed CLL (according to IWCLL guidelines, RMH score 4-5 or RMH 3 providing CD200high and CD20low), excluding small lymphocytic lymphoma without lymphocytosis.
* Indication for treatment according to the 2018 IWCLL criteria and clinically measurable disease.
* Risk stratification: no criteria characterizing low-risk or high-risk groups.
* Patient with unmutated status
* Absence of 17p deletion and/or TP53 mutation.
* Performance status ECOG < 2.
* CIRS (Cumulative Illness Rating Scale) ≤ 6.
* Eligibility for fludarabine, cyclophosphamide and rituximab combination (FCR) and for ibrutinib and venetoclax therapy.
* Adequate hepatic function per local laboratory reference range as follows:
* Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0 x ULN
* Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin).
* No prior treatment for CLL (chemotherapy, radiotherapy, immuno-therapy) except steroids for less than 1 month.
* Willingness to accept highly effective methods of contraception for the duration of therapy and 12 months thereafter.
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at Screening.
* Signed (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

Exclusion Criteria:

* Patients with IGHV mutated (except VH3-21/subset #2) with normal karyotype and/or del 13q without TP53 mutation ie low risk patients.
* Patients del 17p and or TP53 mutation ie high risk patients.
* CLL without active disease according to IWCLL 2008 criteria.
* Known HIV seropositivity.
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:
* Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
* Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
* Active and uncontrolled autoimmune cytopenia, including autoimmune hemolytic anemia (AIHA) (isolated positive DAT is not an exclusion criteria) and idiopathic thrombocytopenic purpura (ITP).
* Life expectancy < 6 months.
* Patient refusal to perform the bone marrow biopsy for evaluation points.
* Active second malignancy currently requiring treatment (except basal cell carcinoma, in situ endometrial carcinoma and incidental prostate carcinoma) and/or less than 5 years CR after breast cancer.
* Concurrent severe diseases which exclude the administration of therapy.
* heart insufficiency NYHA grade III/IV, LEVF < 50% and or RF <30%, myocardial infarction within the past 6 months prior to study.
* severe chronic obstructive lung disease with hypoxemia.
* severe diabetes mellitus.
* hypertension difficult to control.
* impaired renal function with creatinine clearance < 50 ml/min according the formula of Cockcroft and Gault.
* Treatment with any of the following within 7 days prior to the first dose of study drug:
* steroid therapy for anti-neoplastic intent.
* A significant history of renal, neurologic, psychiatric, endocrine, metabolic, immunologic, cardiovascular, or hepatic disease that, in the opinion of the investigator, would adversely affect the patient's participation in this study or interpretation of study outcomes.
* Major surgery within 30 days prior to the first dose of study treatment.
* History of prior other malignancy that could affect compliance with the protocol or interpretation of results, with the exception of the following:
* curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix at any time prior to study.
* other cancers not specified above that have been curatively treated by surgery and/or radiation therapy from which patient is disease-free for ≥ 5 years without further treatment.
* Contraindication to the use of Rituximab.
* Contraindication to the use of Venetoclax.
* Contraindication to the use of Ibrutinib.
* Pregnant or breastfeeding women.
* Adult under law-control.
* Fertile male and female patients who cannot or do not wish to use an effective method of contraception, during and for 12 months after the final treatment used for the purposes of the study.
* No affiliation to social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) in bone marrow (BM) < 0.01% at month 27 | 27 month after beginning FCR or venetoclax + ibrutinib
  MRD evaluation performed by 8 colours flow cytometry analysis in the bone marrow

SECONDARY OUTCOMES:
Progression-free survival (PFS), | from date of inclusion to the date of first-documented progression, assessed up to 4 years
  time from date of randomization to documented progression or death
Complete response (CR) rate at month 9 | at month 9 in the two arms (i.e. 3 months after the 6th cycle of FCR or after 6 months of combined therapy with ibrutinib and venetoclax)
  CR rate (according to IWCLL criteria) with minimal residual disease < 0.01% in bone marrow and undetectable MRD in the blood (with a limit of detection of at least 10-5)
Number of patients with bone marrow MRD < 0.01% at month 9 | At month 9 after beginning FCR or venetoclax + ibrutinib
  Number of patients with MRD < 0.01% by 8 colours flow cytometry analysis in the bone marrow
Complete response (CR) rate at month 27 | at month 27 in the two arms (i.e. 3 months after the 6th cycle of FCR or after 6 months of combined therapy with ibrutinib and venetoclax)
  CR rate (according to IWCLL criteria) with minimal residual disease < 0.01% in bone marrow and undetectable MRD in the blood (with a limit of detection of at least 10-5)
Overall survival (OS) | from date of inclusion to the date of death assessed up to 75 months
  time from date of randomization to date of death or the last date the patient is known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie MICHALLET, Principal Investigator — Centre Leon Berard
Locations (34):
- France (34):
  - CH Annecy Genevois - Hématologie A3, Annecy
  - Ch Cote Basque, Bayonne
  - CH BLOIS, Blois
  - Hôpital Avicenne - Centre de Recherche Clinique, Bobigny
  - Institut Bergonie, Bordeaux
  - CHU Caen - IHBN - Hématologie Clinique, Caen
  - Hôpital Privé Sévigné, Cesson-Sévigné
  - CHU Estaing - Hématologie Clinique Adulte, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Chu Creteil, Créteil
  - GRENOBLE GHM - Institut Daniel Hollard, Grenoble
  - CHU Grenoble - Hématologie, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier du Mans, Le Mans
  - Hôpital Saint Vincent de Paul, Lille
  - Centre Léon Bérard - Hématologie, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre Hospitalier Regional Metz Thionville, Metz
  - Hôpital Saint Eloi, Montpellier
  - CHU Hôtel Dieu - Hématologie Clinique, Nantes
  - CHR ORLEANS - Hématologie, Orléans
  - Hôpital Pitié Salpétrière - Hématologie, Paris
  - Bordeaux Pessac, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie - Hématologie et Thérapie Cellulaire, Poitiers
  - Chu Reims, Reims
  - CHU Pontchaillou - Hématologie Clinique BMT-HC, Rennes
  - Centre Henri Becquerel - Service Hématologie Clinique, Rouen
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital Hautepierre - Hématologie, Strasbourg
  - IUCT ONCOPOLE - Hématologie, Toulouse
  - Hôpital Bretonneau - Hématologie et Thérapie Cellulaire, Tours
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
  - Hôpital André Mignot, Versailles

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the participant data (DPI) collected in this study may be made available to other researchers who request it from the sponsor and if the rationale is the improvement of knowledge in the CLL. The provision will be evaluated by the sponsor.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the end of the study and as long as the sponsor retains the data
Access Criteria: if the rationale is the improvement of knowledge in the CLL